CLINICAL TRIAL: NCT03918200
Title: Serum Amyloid A Level in Women With Unexplained Infertility
Brief Title: Serum Amyloid A in Women With Unexplained Infertility
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Zeinab Saad Abd El Wahab, Doctor, Ain Shams Maternity Hospital
Other Study IDs: SAAI
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study: Women with unexplained infertility
  Interventions: Other: Serum amyloid A level
- Control: Fertile women who had normal physical and pelvic examination, regular menstrual cycles, don't use hormonal contraceptive, had one child at least.
  Interventions: Other: Serum amyloid A level

INTERVENTIONS:
Other: Serum amyloid A level — For determination of SAA level, a 5-ml sample of venous blood will be taken from each participant under aseptic conditions, and centrifuged at 2500 g for 15 minutes at 4°C c. separated into serum aliquots,and stored frozen at -80°C until analysis of SAA ,which will be done by a double-antibody sandwich Enzyme Linked Immunosorbent Assay (ELISA) kits supplied by cusabio,USA according to manufacturers instruction .Each sample was tested in duplicate and the average will be taken. A cut off level of 30 mg/L SAA level will be chosen to reflect a real increase in its level

SUMMARY:
High follicular fluid amyloid A level is associated with reduced pregnancy rate.

The aim of this study was to find an association between serum level of amyloid A and unexplained infertility.

ELIGIBILITY:
Inclusion Criteria:

1. women with unexplained infertility (unprotected, regular intercourse for at least 2 years).
2. Nulligravida ,Regular mensturation.
3. Age less than 40 years .
4. Normal parameters (in the study group):

   * hormonal profile (day 2 FSH,LH), midluteal phase progesterone, Prolactin, TSH
   * transvaginal ultrasound
   * hysterosalpingography
   * detailed semen analysis

Exclusion Criteria:

1. Age above 40
2. Smoking females
3. Obesity (BMI>30)
4. Women with any systemic or medical diseases leads to elevation of SAA as:

   1. Systemic lupus erythematosis
   2. Rheumatoid arthritis
   3. Sarcoidosis
   4. Diabetes Mellitus
5. Using hormonal contraception (for control group)

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Infertile women attending Ain Shams University infertility outpatient clinic seeking fertility and fulfilling the criteria.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Difference between SAA level between cases and control. | 1 day (once)

SECONDARY OUTCOMES:
Correlation between SAA level with other parameters in the hormonal profile (e.g., FSH, LH, E2). | 1 day (once)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided